CLINICAL TRIAL: NCT05852925
Title: Evaluation of Tasso+ Capillary Blood Self-Collection for Clinical Diagnostic Assessment of Various Biomarkers
Brief Title: Evaluation of Tasso+ Blood Self-Collection for Clinical Diagnostic Assessment of Various Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Research Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00069812
Record Dates: First submitted 2023-03-14; First posted 2023-05-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Blood Self-Collection for Clinical Diagnostic Assessments

STUDY DESIGN:
Intervention Model Description: The study is an interventional single-group model, using a single-arm design in which all participants receive the same interventions, which includes the traditional venipuncture and Tasso+ blood self-collection. Both collection procedures are performed sequentially at the study site, with a phlebotomist performing the traditional venipuncture followed by the participant collecting blood using the Tasso+ device following provided instructions independently. The lab results will be analyzed to assess the correlation of biomarkers between blood samples obtained using the Tasso+ device and those collected via venipuncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Human Blood Specimen Collection (Other): Blood will be collected from each participant using two different methods: the Tasso+ device and the traditional venipuncture approach. Both collection procedures are carried out sequentially at the study site. A phlebotomist performs the traditional venipuncture and the participant collects blood using two Tasso+ devices, following provided instructions. The lab results will be analyzed to assess the correlation of biomarkers between blood samples obtained by the participant using the Tasso+ device and those collected via venipuncture.
  Interventions: Other: Traditional Venipuncture; Device: Tasso+

INTERVENTIONS:
Other: Traditional Venipuncture — Traditional blood collection is performed and the necessary amount of blood is collected into the collection tubes (either SST or Lithium Heparin tubes based on the biomarker being tested).
Device: Tasso+ — The Tasso+ is the blood self-collection device used in the study and this device enables the collection of microliter capillary whole blood samples into compatible reservoirs. In this study, the reservoirs utilized include either SST or Lithium Heparin microtainers based on the biomarker being tested.

SUMMARY:
This study aims to assess the effectiveness and reliability of the Tasso+ capillary blood self-collection device in the clinical diagnostic assessment of various biomarkers. The study will collect blood specimens using both the Tasso+ self-collection device and traditional venipuncture. The biomarker analysis results from both specimen types will be compared for correlation.

DETAILED DESCRIPTION:
A kit containing all required supplies for traditional blood collection as well as Tasso+ self-collection kits for blood will be provided to the study sites. The kit will also include any additional supplies necessary for the collection process. The complete kit will be shipped to the sites as a single unit.

1. Research staff will approach subjects to determine their interest in participating in this study that involves both traditional venipuncture and Tasso+ blood self-collection procedures. If a subject is willing, a qualified study team member will obtain their agreement, conduct the informed consent process, document the participant's consent, and provide them with a copy of the informed consent form information sheet.
2. Study staff will complete the necessary source document elements and case report forms, collecting relevant subject demographic information, eligibility criteria, and medical history. Blood will be collected from each participant using two different methods: the Tasso+ device and the traditional venipuncture approach. Both collection procedures are carried out sequentially at the study site. A phlebotomist performs the traditional venipuncture followed by the participant collecting blood using the Tasso+ device following the provided instructions independently. The lab results will be analyzed to assess the correlation of biomarkers between blood samples obtained by the participant using the Tasso+ device and those collected via venipuncture.
3. The analysis will focus on the potential biomarkers as listed. Albumin, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Alpha-Fetoprotein (AFP), Anti-CCP (Cyclic citrullinated peptide), Thyroglobulin antibody (Anti-Tg), Thyroid Peroxidase Antibodies (Anti-TPO), Aspartate Aminotransferase (AST), Bilirubin Direct, Bilirubin Total, BUN Serum, Cancer Antigen (CA) 125, Cancer Antigen (CA) 15-3, Carbohydrate Antigen (CA) 19-9 XR, Calcium, Cancer Antigen (CA) 15-3, Carcinoembryonic antigen (CEA), Cholesterol Total, Chloride, Carbon Dioxide Total, Cortisol, C-Reactive Protein (CRP) Cardiac, C-Reactive Protein (CRP) Wide range, C-Reactive Protein High sensitivity (CRPHS), Creatinine Serum, Low-density Lipoprotein Cholesterol (Direct LDL), Dehydroepiandrosterone (DHEA), Dehydroepiandrosterone Sulfate (DHEA-S) , Estradiol, Ferritin, Folate, Thyroxine(T4) Free, Triiodothyronine (T3) Free, Follicle-stimulating Hormone (FSH), Globulin Total, Glucose, Growth Hormone, Hemoglobin A1c (HbA1c), High-density Lipoprotein (HDL) Cholesterol, Hepatitis A Antibody IgM, Hepatitis B Core Antibody IgM, Hepatitis B Surface Antigen (HBsAg) Screen, Hepatitis B Surface Antigen (HBsAg) Confirmatory, Hepatitis C Virus (HCV) Antibody, HIV Antigen/ Antibody Combo, Herpes I & II IgG, Iron, Luteinizing Hormone (LH), Mumps Antibodies IgG, Potassium, Progesterone, Prolactin, Protein Total, Rheumatoid Factor (RF), Rubella IgG Antibodies, Rubella IgM Antibodies, Rubeola Antibodies IgG, Sodium, Treponema pallidum Antibodies (Syphilis), Testosterone Free, Testosterone Total, Thyroxine(T4), Total Iron-binding Capacity (TIBC), Triiodothyronine (T3), Triglycerides, Thyroid-stimulating Hormone (TSH), Varicella IgG antibodies, Vitamin B12, Vitamin D 25-Hydroxy, PSA Total, Human Chorionic Gonadotropin (β-hCG) Qualitative, Human Chorionic Gonadotropin (β-hCG) Quantitative, Sex hormone binding globulin (SHBG), Apolipoprotein B(ApoB), Lipoprotein(a) [Lp(a)], Glial fibrillary acidic protein (GFAP), Ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1), Complete Blood Count with Differential, CBC. In addition to the biomarkers listed, the protocol will encompass the testing of additional potential biomarkers not listed, to allow for the exploration of new analytes as they become clinically relevant. The biomarkers are quantified or qualitatively measured using either Abbott Alinity ci-series, Siemens Dimension EXL, Siemens Immulite 200 xpi, Dynex DSX Automated Elisa System or an equivalent analyzer. Note: A biomarker collected from both venipuncture and Tasso+ methods will be analyzed using the same analyzer to avoid any bias that may arise from using different instruments.
4. Traditional blood collection is performed, and the necessary amount of blood is drawn into the collection tubes. The type of tube used, either SST or Lithium Heparin, depends on the specific biomarker being tested in the study.
5. The Tasso+ is the blood self-collection device used in the study and this device enables the collection of microliter capillary whole blood samples into compatible reservoirs. In this study, the reservoirs utilized will be either SST microtainer or Lithium Heparin microtainer. A subject collects blood using two Tasso+ devices, selecting either the SST microtainer or the Lithium heparin microtainer based on the specific biomarker being tested in the study.
6. The subject receives a Tasso+ blood collection kit, which includes a Tasso+ device, a biohazard bag, an alcohol swab, and an instruction manual. The subject should read and follow the instruction manual which includes steps for at-home kit registration, blood self-collection process, packaging, and shipping guidelines.
7. Participation in this trial is not expected to provide any potential benefits to the subject. However, the knowledge gained could potentially contribute to the future adoption of the Tasso+ device for safe, at-home blood self-collection. The study simulates remote home collection by having subjects follow the instructions and perform the blood self-collection independently using the Tasso+ device.
8. Blood collected in traditional venipuncture tubes (SST and Lithium Heparin) will be centrifuged, while Tasso+ samples collected in SST and Lithium Heparin microtainers will not undergo centrifugation. Tasso+ samples are not centrifuged to mimic at-home patient testing, where patients do not centrifuge the sample before shipping. These Tasso+ samples will be centrifuged at the laboratory. However, for sample equivalence studies, the study staff will centrifuge a subset of Tasso+ samples. Both traditional venipuncture and Tasso+ self-collection samples will be sent to the laboratory to perform clinical diagnostic testing for the biomarkers.
9. The lab results will be analyzed to assess the correlation of biomarkers between blood samples obtained using the Tasso+ device and those collected via venipuncture. The diagnostic results of biomarkers will be compared between traditional venipuncture and Tasso+ self-collection methods, and reference intervals for the biomarkers collected using the Tasso+ self-collection device will be established as needed.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, an individual must meet all the following criteria:

1. Age: Participants must be 13 years of age or older.
2. Medical history: There may be no specific medical history requirements for inclusion, although participants may need to meet certain general health criteria.
3. Sample type: Participants must be willing and able to provide the human specimens needed for the study, such as blood, urine, or saliva.
4. Ability to provide consent: Participants must have the ability to provide informed consent to participate in the study, either on their own behalf if they are legally able to do so, or with the consent of a parent or guardian if they are under 18 years of age.
5. Language proficiency: Participants must be able to read and understand the language used in the study materials, such as informed consent forms and instructions for specimen collection.

Exclusion Criteria:

Participation in this study will be excluded for individuals who meet the following criterion:

1. Blind or visually impaired: Participants who are unable to see or have significant visual impairment that would make it difficult for them to participate in the study.
2. Decisionally impaired: Participants who are unable to provide informed consent due to cognitive impairment, developmental disability, or other mental health conditions that affect decision-making capacity.
3. Educationally disadvantaged: Participants who lack the education or literacy skills required to understand the study procedures or provide informed consent.
4. Hospitalized: Participants who are currently hospitalized, as they may not be able to participate in the study due to their medical condition or limited mobility.
5. Prisoners: Participants who are incarcerated in correctional facilities, as their participation may raise ethical concerns or require additional regulatory approvals.
6. Terminally ill: Participants who have a terminal illness or life-limiting condition that may affect the study results or pose additional risks to their health.

Excluding individuals with these characteristics from the study is intended to ensure their safety and well-being and to maintain the integrity of the study results.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Venous and Tasso+ blood sample correlation for biomarkers being tested. | 1 Year
  Correlation between the venous blood sample with the Tasso+ blood sample for the biomarkers listed in the study description.
  The biomarkers are quantified or qualitatively measured using either Abbott Alinity ci-series, Siemens Dimension EXL, Siemens Immulite 2000 xpi, Dynex DSX Automated Elisa System, or an equivalent analyzer.
  Note: A biomarker collected from both venipuncture and Tasso+ methods will be analyzed using the same analyzer to avoid any bias that may arise from using different instruments

SECONDARY OUTCOMES:
Collect patient experience with the Tasso+ blood collection device kit. | 1 Year
  A brief survey will be designed to understand the subject's experience with the Tasso+ blood collection device kit to perform independent kit registration, independent sample collection, and packaging to simulate remote self-collection.

CONTACTS AND LOCATIONS:
Overall Officials: Sri Bharat Madireddy, Ph.D., Principal Investigator — American Research Labs; Vanaja Reddy Bodeddula, Ph.D., Study Director — American Research Labs
Locations (1):
- American Research Labs, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No